CLINICAL TRIAL: NCT06248892
Title: A Randomized Controlled Study to Explore the Clinical The Effect of Oral and Nasal Feeding on Cerebral Small Vessel Disease
Brief Title: The Effect of Oral and Nasal Feeding on Cerebral Small Vessel Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zeng Changhao (Other)
Responsible Party: Sponsor-Investigator, Zeng Changhao, Research Director, People's Hospital of Zhengzhou University
Organization: People's Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IOE-CVSD new
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Cerebral Small Vessel Diseases
MeSH Terms: conditions — Cerebral Small Vessel Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The observation group (Experimental): Assigned by the random number table. During the treatment, all patients were provided with comprehensive rehabilitation therapy.
  Besides, the observation group was given enteral nutritional support with Intermittent Oro-esophageal Tube Feeding according to the relevant guidelines.
  Interventions: Device: Intermittent Oro-esophageal Tube Feeding; Behavioral: comprehensive rehabilitation therapy
- The control group (Active Comparator): Assigned by the random number table. During the treatment, all patients were provided with comprehensive rehabilitation therapy.
  Besides, the control group was given enteral nutritional support with nasogastric tube according to the relevant guidelines. Within 4 hours after admission, the placement of the feeding tube was conducted by professional medical staffs and after intubation.
  Interventions: Device: Nasogastric Tube Feeding; Behavioral: comprehensive rehabilitation therapy

INTERVENTIONS:
Device: Nasogastric Tube Feeding — Nasogastric Tube Feeding were used for feeding to provide nutritional support. Each feeding was administered by a nurse using the infant's mother's breast milk through the tube. The amount of each feeding varied from 20 to 100 ml depending on the age of the infant, with feedings given every 2 to 3 hours, approximately 10 times per day. The duration of each feeding procedure ranged from 10 to 20 minutes. The total daily intake ranged from 200 to 1000 ml. Each tube was kept indwelling for 5 to 7 days. When the tube needed to be replaced, it was removed after the last feeding of a day and a new tube was to be inserted through the other nostril on the following morning to continue the nutritional support.
  Arms: The control group
Device: Intermittent Oro-esophageal Tube Feeding — The specific procedure was as follows: the infant was placed in a semi-recumbent or sitting position with the head fixed. Before each feeding, the infant's oral and nasal secretions were to be cleared. An intermittent oro-esophageal tube was appropriately lubricated with water on the head part. The professional medical staff held the tube and slowly inserted it through one side of the mouth into the upper part of the esophagus. The depth of insertion depended on the patient's age and height. After each feeding, the tube was immediately removed, and the patient was held upright for at least 30 minutes in case of reflux.
  Arms: The observation group
Behavioral: comprehensive rehabilitation therapy — Both groups were given comprehensive rehabilitation therapy. The main intervention measures included: 1) non-invasive ventilator treatment, generally at least once every night and typically not exceeding continuous daily usage.; 2) attention to feeding and sleeping positions, with a recommended sleeping position of lateral recumbent and the head of the bed raised by 20-30°; 3) swallowing function training, such as tongue muscle stretching training, assisted anterior jaw protrusion training, lemon ice stimulation to the soft palate, pharyngeal wall, etc., generally 5 days per week, twice per day, 5-20 minutes each time; 4) pulmonary ultrashort wave therapy, generally at least 2-3 times a week, and not more than once a day; 5) physical therapy, such as intensive training for gross motor functions including lifting the head, turning over, sitting, crawling, standing, etc., generally 3-5 days per week, 1-2 times per day, 5-20 min each time.

SUMMARY:
Nasogastric tube feeding (NGT) has been widely used in cerebral small vessel disease (CSVD) patients with dysphagia but has a significant risk of complications. Intermittent Oro-esophageal Tube Feeding (IOE) is an established enteral nutrition approach that can be used with comprehensive rehabilitation therapy. This study aims to explore the clinical effect of IOE vs. NGT on CSVD Patients with Dysphagia. Compared to NGT, IOE, as an enteral nutrition support mode, in CSVD Patients with Dysphagia who received comprehensive rehabilitation therapy, showed advantages in improvement in dysphagia, nutritional status, ADL, QOL, pneumonia, and adverse events, which should be considered as the preferred approach.

DETAILED DESCRIPTION:
Nasogastric tube feeding (NGT) has been widely used in cerebral small vessel disease (CSVD) patients with dysphagia but has a significant risk of complications. Intermittent Oro-esophageal Tube Feeding (IOE) is an established enteral nutrition approach that can be used with comprehensive rehabilitation therapy. This study aims to explore the clinical effect of IOE vs. NGT on CSVD Patients with Dysphagia.

This was a randomized controlled study with 60 CSVD Patients with Dysphagia who received comprehensive rehabilitation therapy. Patients enrolled were randomly divided into the observation group (with IOE, n=30) and the control group (with NGT, n=30). At admission and after treatment, Video Fluoroscopic Swallowing Study (VFSS) and Functional Oral Intake Scale (FOIS), body mass index (BMI), serum albumin (Alb), and hemoglobin (Hb), Modified Barthel Index (MBI) and World Health Organization Quality of Life Assessment Instrument Brief Version (WHOQOL-BREF) were recruited to assess and compare dysphagia, nutritional status, activities of daily living (ADL) and quality of life (QOL). The incidence of pneumonia was recorded and compared.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Cerebral Small Vessel Disease;
* Must be able to cooperate with treatment and questionnaire investigation, (Generally with a Mini-Mental State Examination (MMSE) score ≥ 24) ;
* Clinical diagnosis of dysphagia through the Functional Oral Intake Scale (FOIS) and Video Fluoroscopic Swallowing Study (VFSS);
* Age between 40 and 70 years;
* Enteral nutrition support was required and feasible.
* No history of prior stroke.

Exclusion Criteria:

* Dysphagia related to other cerebrovascular diseases or caused by neurodegenerative diseases;
* Complicated with severe liver and kidney failure, tumors, or hematological disorders;
* Simultaneously need to undergo other therapy that might affect the outcomes of this study;
* Pregnant or nursing females.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Video Fluoroscopic Swallowing Study | day 1 and day 15
  Video Fluoroscopic Swallowing Study, which is considered as the "gold standard", swallowing process is divided into four periods: cognitive, oral, pharyngeal, and esophageal periods with a total score of 10 and a higher score indicates better swallowing ability (less dysphagia).

SECONDARY OUTCOMES:
Functional Oral Intake Scale | day 1 and day 15
  During Dysphagia-Functional Oral Intake Scale assessment, evaluators engage in communication with the patient, conduct observations, and make records to assess the patient's oral intake ability. The FOIS assessment form includes seven levels of scoring, ranging from level 1 to level 7, indicating a progressive improvement in the patient's oral intake ability. In general, the result below level 6 indicates unsafe for oral intake while level 6 and above indicates that eating via mouth can be safely conducted.
Body mass index | day 1 and day 15
  Weight and height will be combined to report Body mass index in kg/m^2
Serum albumin | day 1 and day 15
  Serum albumin was recorded via blood routine test.(Alb, g/L)
Hemoglobin | day 1 and day 15
  Hemoglobin was recorded via blood routine test.(Hb, mg/L)
Pneumonia | day 1 and day 15
  The occurrence of pneumonia in patients was assessed before and after treatment. Specifically, first of all, the symptom assessment and physical examination were conducted to all patients, during which, the doctor would inquire symptoms related to pneumonia, such as cough, sputum production, difficulty breathing, chest pain, etc. and observe the patient's respiratory condition, including respiratory rate, breath sounds, and any abnormal signs in the chest. If there was probability for potential pneumonia, patients were requested for further diagnosis
Activities of daily living | day 1 and day 15
  The activities of daily living was assessed utilizing the Modified Barthel Index (MBI). Modified Barthel Index includes the following 10 subscales. For each subscale, choices encoded with the score 10, 8, 5, 2, 0 are set with the decreasing level of self-dependence, while the final total is positively correlated with Activities of daily living. Cronbach's α of questionnaire adopted is 0.916.
World Health Organization Quality of Life Assessment Instrument Brief Version | day 1 and day 15
  The Quality of Life was assessed utilizing the World Health Organization Quality of Life Assessment Instrument Brief Version (WHOQOL-BREF). WHOQOL-BREF covers various aspects such as mobility, pain, emotions, personal relationships, living conditions, and access to health services, to evaluate Quality of Life. Each item is rated on a Likert scale, and the scores are transformed into a standardized score ranging from 0 to 100, with higher scores indicating better Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Principal Investigator — Site Coordinator of United Medical Group located in Miami
Locations (1):
- Ratchaburi Center Hos., Ratchaburi, Thailand

IPD SHARING:
Plan to Share IPD: No